CLINICAL TRIAL: NCT06741878
Title: A Biopsychosocial Approach to Improving Multidimensional Frailty Status in Community-Dwelling Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Baptist University (Other)
Collaborators: Coburg University of Applied Sciences and Arts (Unknown); The Hong Kong Polytechnic University (Other); Tung Wah College (Other); Research Grants Council, Hong Kong (Other); Constructor University (Unknown)
Responsible Party: Principal Investigator, JIAO Jiao, Research Assistant Professor, Hong Kong Baptist University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 12600824
Record Dates: First submitted 2024-12-11; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Frailty in Older Adults
Keywords: Multi-dimensional frailty; Biopsychosocial approach; Exercise training; Nutrition education; Psychosocial support; Older adults; Intervention programs
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Exercise Training (Biological) + Board Games (Psychosocial) + Diet Consultation (Nutritional) (Active Comparator)
  Interventions: Behavioral: Exercise; Behavioral: Psychosocial; Behavioral: Nutritional
- Exercise Training (Biological) + Diet Consultation (Nutritional) (Active Comparator)
  Interventions: Behavioral: Exercise; Behavioral: Nutritional
- Board Games (Psychosocial) + Diet Consultation (Nutritional) (Active Comparator)
  Interventions: Behavioral: Psychosocial; Behavioral: Nutritional
- Inactive Control (No Treatment) (No Intervention)

INTERVENTIONS:
Behavioral: Exercise — Involves participants engaging in physical training group sessions in light-to-moderate intensity.
  Arms: Exercise Training (Biological) + Board Games (Psychosocial) + Diet Consultation (Nutritional); Exercise Training (Biological) + Diet Consultation (Nutritional)
Behavioral: Psychosocial — Involves participants engaging in selected board and card games which require cognitive and socialization skills to play in a group setting of 2-4 people.
  Arms: Board Games (Psychosocial) + Diet Consultation (Nutritional); Exercise Training (Biological) + Board Games (Psychosocial) + Diet Consultation (Nutritional)
Behavioral: Nutritional — Involves participants attending dietary classes taught by a certified dietitian, including individualized consultation.
  Arms: Board Games (Psychosocial) + Diet Consultation (Nutritional); Exercise Training (Biological) + Board Games (Psychosocial) + Diet Consultation (Nutritional); Exercise Training (Biological) + Diet Consultation (Nutritional)

SUMMARY:
Frailty is a common clinical syndrome that is becoming increasingly important as populations age worldwide. Individuals who are frail are at a higher risk for negative outcomes, such as falls, disability, hospitalizations, and even death. The understanding of frailty has evolved from a straightforward concept to a complex model that includes physical, psychological, cognitive, and social factors. Since frailty is not static and can change over time, early interventions can be beneficial. Nevertheless, research in this area has been challenging due to a lack of agreement on what frailty encompasses and an inadequate understanding of how its different components interact. Defining frailty as a multidimensional issue is essential to recognize the adverse effects that can arise from medical, psychological, and social influences. However, recent studies have not sufficiently addressed how these different aspects work together or developed effective multidimensional interventions.

DETAILED DESCRIPTION:
The study will be designed as a four-arm, double-blinded, cluster-randomised controlled trial. A sample (N = 308) of prefrail older adults aged 60-80 years will be recruited from 32 randomly selected elderly community centres in Hong Kong and classified into four frailty deficit patterns (multi-frailty, physical-to-psycho/social, nonphysical-to-psycho/social, and a robust control). With the hypothesised biopsychosocial framework pinpointing the intertwined relationships of these three domains of frailty, four intervention strategies (biological/psychosocial/nutritional, biological/nutritional, psychosocial/nutritional, and an inactive control) will be proposed to improve their overall frailty, regarding their physical, psychological, and social functioning, nutritional status, and lifestyle changes in a 9-month intervention and follow-up period. The primary objective will be to assess the effectiveness of the intervention strategies for improving the frailty status of participants in each of the four frailty deficit pattern groups, and to determine the most effective intervention strategy.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 to 80
* Willing and capable to participate in this study and training
* Willing and capable to give informed consent to participate in this study
* Preliminarily classified as physically prefrail/robust, in that they possess no more than three of the indicators on the Fried Frailty Index (FFI; unintentional weight loss, exhaustion, low physical activity, slow walking speed, weak grip strength; Bieniek et al., 2016)
* Can walk independently to an elderly centre
* Have a smartphone for internal group communication and remote interaction with their peers and the instructor

Exclusion Criteria:

* History of systematic cardiovascular diseases causing stroke, Parkinson's disease, early stages of Alzheimer's disease, or cognitive impairment
* Physical injuries or other conditions that would hinder regular attendance and participation in the assessments for the study
* Concurrent major psychiatric disorder (e.g. major depressive disorder, schizophrenia) or drug and alcohol abuse
* Unable to handle digital devices
* Currently undergoing exercise programmes or classified as physically 'very active' (i.e. performing strenuous activity for 5+ hours each week)

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 308 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Frailty Status (pre-test) | Pre-test (1st test): before intervention
  The Tilburg Frailty Indicator (TFI), with three subdomains (physical, psychological, and social), will be used in three evaluation time frames, respectively. The total TFI score ranges from 0 to 15, with a score of 5 (or above) indicating frailty.
Frailty Status (2nd test) | 2nd test: after 3-month intervention
  The Tilburg Frailty Indicator (TFI), with three subdomains (physical, psychological, and social), will be used in three evaluation time frames, respectively. The total TFI score ranges from 0 to 15, with a score of 5 (or above) indicating frailty.
Frailty Status (3rd test) | 3rd test: after 6-month follow up
  The Tilburg Frailty Indicator (TFI), with three subdomains (physical, psychological, and social), will be used in three evaluation time frames, respectively. The total TFI score ranges from 0 to 15, with a score of 5 (or above) indicating frailty.
Physical Functioning-- Anthropometic Data (pre-test) | Pre-test (1st test): before intervention
  Anthropometric data (e.g. BMI in kg/m^2) will be evaluated in 3 time frames, respectively.
Physical Functioning-- Anthropometric Data (2nd test) | 2nd test: after 3-month intervention
  Anthropometric data (e.g. BMI in kg/m^2) will be evaluated in 3 time frames, respectively.
Physical Functioning-- Anthropometric Data (3rd test) | 3rd test: after 6-month follow up
  Anthropometric data (e.g. BMI in kg/m^2) will be evaluated in 3 time frames, respectively.
Physical Functioning-- Health Related Information (pre-test) | Pre-test (1st test): before intervention
  Health-related information (heart rate, daily step counts, etc.) collected by a Smart Band will be used in three evaluation time frames, respectively.
Physical Functioning-- Health Related Information (2nd test) | 2nd test: after 3-month intervention
  Health-related information (heart rate, daily step counts, etc.) collected by a Smart Band will be used in three evaluation time frames, respectively.
Physical Functioning-- Health Related Information (3rd test) | 3rd test: after 6-month follow up
  Health-related information (heart rate, daily step counts, etc.) collected by a Smart Band will be used in three evaluation time frames, respectively.
Physical Functioning-- Senior Physical Fitness Test Battery (pre-test) | Pre-test (1st test): before intervention
  The senior physical fitness test battery (SPFT) (Jones, 2013) will be used in three evaluation time frames, respectively. The SPFT consists of six physical tests for assessing functional fitness in the elderly: 30 sec arm curl (muscular strength), 30 sec chair stand (muscular strength), 2 min step test (aerobic endurance), chair sit-and-reach (flexibility), back scratch test (flexibility), and up-and-go (dynamic balance).
Physical Functioning-- Senior Physical Fitness Test Battery (2nd test) | 2nd test: after 3-month intervention
  The senior physical fitness test battery (SPFT) (Jones, 2013) will be used in three evaluation time frames, respectively. The SPFT consists of six physical tests for assessing functional fitness in the elderly: 30 sec arm curl (muscular strength), 30 sec chair stand (muscular strength), 2 min step test (aerobic endurance), chair sit-and-reach (flexibility), back scratch test (flexibility), and up-and-go (dynamic balance).
Physical Functioning-- Senior Physical Fitness Test Battery (3rd test) | 3rd test: after 6-month follow up
  The senior physical fitness test battery (SPFT) (Jones, 2013) will be used in three evaluation time frames, respectively. The SPFT consists of six physical tests for assessing functional fitness in the elderly: 30 sec arm curl (muscular strength), 30 sec chair stand (muscular strength), 2 min step test (aerobic endurance), chair sit-and-reach (flexibility), back scratch test (flexibility), and up-and-go (dynamic balance).
Psychological Functioning (pre-test) | Pre-test (1st test): before intervention
  A seven-item scale of psychological well-being, which is an indicator of psychological functioning in the Comprehensive Model of Frailty (CMF) (Kwan et al., 2015), will be used in three evaluation time frames, respectively.
Psychological Functioning (2nd test) | 2nd test: after 3-month intervention
  A seven-item scale of psychological well-being, which is an indicator of psychological functioning in the Comprehensive Model of Frailty (CMF) (Kwan et al., 2015), will be used in three evaluation time frames, respectively.
Psychological Functioning (3rd test) | 3rd test: after 6-month follow up
  A seven-item scale of psychological well-being, which is an indicator of psychological functioning in the Comprehensive Model of Frailty (CMF) (Kwan et al., 2015), will be used in three evaluation time frames, respectively.
Social Function (pre-test) | Pre-test (1st test): before intervention
  The risk of social functioning deficits will be tested using the Social Frailty Index (SFI) in three evaluation time frames, respectively.
Social Function (2nd test) | 2nd test: after 3-month intervention
  The risk of social functioning deficits will be tested using the Social Frailty Index (SFI) in three evaluation time frames, respectively.
Social Function (3rd test) | 3rd test: after 6-month follow up
  The risk of social functioning deficits will be tested using the Social Frailty Index (SFI) in three evaluation time frames, respectively.

SECONDARY OUTCOMES:
Physical Activity Behavioural Changes (pre-test) | Pre-test (1st test): before intervention
  Scales of physical activity behavioural change, intention/motivation, loneliness, subjective physical health, and health status will be measured using a survey that was used in a previous project (Chow et al., 2022), in three time frames.
Physical Activity Behavioural Changes (2nd test) | 2nd test: after 3-month intervention
  Scales of physical activity behavioural change, intention/motivation, loneliness, subjective physical health, and health status will be measured using a survey that was used in a previous project (Chow et al., 2022), in three time frames.
Physical Activity Behavioural Changes (3rd test) | 3rd test: after 6-month follow up
  Scales of physical activity behavioural change, intention/motivation, loneliness, subjective physical health, and health status will be measured using a survey that was used in a previous project (Chow et al., 2022), in three time frames.
Exercise Self-efficacy (pre-test) | Pre-test (1st test): before intervention
  Assessed using the validated Chinese scales of the Physical Exercise Self-efficacy Scale (PESES), a 5-item instrument with a 4-point Likert-type scale, ranging from 5 to 20. Higher scores shows higher routine physical exercise self-efficacy.
Exercise Self-efficacy (2nd test) | 2nd test: after 3-month intervention
  Assessed using the validated Chinese scales of the Physical Exercise Self-efficacy Scale (PESES), a 5-item instrument with a 4-point Likert-type scale, ranging from 5 to 20. Higher scores shows higher routine physical exercise self-efficacy.
Exercise Self-efficacy (3rd test) | 3rd test: after 6-month follow up
  Assessed using the validated Chinese scales of the Physical Exercise Self-efficacy Scale (PESES), a 5-item instrument with a 4-point Likert-type scale, ranging from 5 to 20. Higher scores shows higher routine physical exercise self-efficacy.
Nutrition Self-efficacy (pre-test) | Pre-test (1st test): before intervention
  Assessed using the Nutrition Self-efficacy Scale (NSES) (Schwarzer, 2009; Wong et al., 2020).
Nutrition Self-efficacy (2nd test) | 2nd test: after 3-month intervention
  Assessed using the Nutrition Self-efficacy Scale (NSES) (Schwarzer, 2009; Wong et al., 2020).
Nutrition Self-efficacy (3rd test) | 3rd test: after 6-month follow up
  Assessed using the Nutrition Self-efficacy Scale (NSES) (Schwarzer, 2009; Wong et al., 2020).
Nutritional Status (pre-test) | Pre-test (1st test): before intervention
  Assessed by the Mini Nutritional Assessment scale (MNA). The MNA score ranges from 0 to 14, with a higher score indicating better nutritional status.
Nutritional Status (2nd test) | 2nd test: after 3-month intervention
  Assessed by the Mini Nutritional Assessment scale (MNA). The MNA score ranges from 0 to 14, with a higher score indicating better nutritional status.
Nutritional Status (3rd test) | 3rd test: after 6-month follow up
  Assessed by the Mini Nutritional Assessment scale (MNA). The MNA score ranges from 0 to 14, with a higher score indicating better nutritional status.

IPD SHARING:
Plan to Share IPD: No
In the application of university human ethics, the investigators have declared non-disclosure of individual data.

REFERENCES:
- [Derived] Jiao J, Man DW, Lippke S, Hassel H, Tam BT, Chan CH, Ng YL, Lo KK. A biopsychosocial approach to improving multidimensional frailty status in community-dwelling older adults: a protocol for a cluster randomized controlled trial. BMC Geriatr. 2025 Jul 15;25(1):530. doi: 10.1186/s12877-025-06053-x. PMID 40665217